CLINICAL TRIAL: NCT02118233
Title: Cognitive Outcome After Carotid Surgery
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-009
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2018-03

CONDITIONS: Carotid Stenosis
Keywords: carotid; stenosis; surgery; cognitive; unilateral
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Carotid Endarterectomy (CEA): Surgical Revascularization- Carotid Endarterectomy (CEA)
- Carotid Angioplasty and Stenting (CAS): Surgical Revascularization- Carotid Angioplasty and Stenting (CAS)
- Control Group- Medical Management: Control Group- Medical Management

SUMMARY:
The purpose of this study is to understand how carotid endarterectomy (CEA) or percutaneous carotid angioplasty and stenting (CAS) affect memory and thinking resulting in improving or worsening of thinking or memory. There have been many studies on this subject, some finding that certain patients gain improvement in their brain function and others might get worse. The goal of this study is to discover which patients are more likely to have improved cognitive functioning. Carotid endarterectomy (CEA) and percutaneous carotid angioplasty and stenting (CAS) are not investigational and are an accepted treatment for your condition. In addition, subjects that choose not to undergo surgery will also be included in this study.

DETAILED DESCRIPTION:
At the present time, large multi-center clinical trials support the use of carotid revascularization for symptomatic carotid stenosis and for asymptomatic carotid stenosis (greater than 60%) to prevent stroke. Guidelines supporting the use of carotid endarterectomy for asymptomatic stenosis are based largely on the Asymptomatic Carotid Atherosclerosis Study (ACAS) which reported a 47% relative risk reduction for ipsilateral stroke or death in patients randomized to surgery compared to best medical management over 5 years. These data were further substantiated by the recent publication of the Medical Research Council Asymptomatic Carotid Surgery (ACST) trial results (1); however, both trials estimated that at least 40 operative procedures were required to prevent a single disabling stroke or death in one patient after 5 years (2). These data underscore the importance of understanding the cognitive risks of carotid revascularization and developing strategies to limit factors that contribute to this risk especially in asymptomatic patients.

The purpose of this study is to better understand the effect of carotid revascularization (using either carotid endarterectomy (CEA) or percutaneous carotid angioplasty and stenting (CAS)) on cognitive outcome by prospectively collecting cerebral blood flow data and cognitive testing data prior to and after carotid revascularization procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asymptomatic (defined as no symptoms in past 6 months) carotid stenosis
* Patients with hemodynamically significant carotid artery stenosis (according to CREST criteria: ≥ 60% by angiography, OR ≥ 70% by ultrasound, OR ≥ 80% by CTA or MRA)

Exclusion Criteria:

* Patients with prior large vessel infarct
* Patients with intracranial stenosis
* Patients with major depression
* Patients with Alzheimer disease (clinically defined or Wechsler IQ <80)
* Patients who have had previous ipsilateral carotid surgery
* Patients with baseline dementia defined as: Mini-Mental Status Examination score < 21 OR Mini-Mental score ≥21 AND Baseline HVLT scores more than 3 standard deviations below normal or FAS scores more than 2 standard deviations below normal OR other clinical symptoms that were not as evident on direct cognitive assessment (e.g. sundowning, getting lost while driving).

Note: A control group would be comprised of about 15 patients who meet eligibility criteria as above, but elect to have their condition followed rather than undergo revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral, asymptomatic, significant carotid artery stenosis who are ≥18 years of age who do not present with past or current significant cerebrovascular and neuropsychological disease.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Measurement of change in cerebral blood flow from pre-op/baseline to 1 month post-operatively. | preoperative/baseline and 1 month postoperative/from baseline
  Quantitative flow MRA studies will be performed pre-operative and postoperative for those undergoing carotid revascularization surgery. Those not undergoing surgery will have this test upon study enrollment and approximately 1 month from study enrollment date.

SECONDARY OUTCOMES:
Mini Mental Status Exam | Pre-operative/baseline
  A standardized cognitive measure
Trail Making- Part A | Preoperative/baseline, 1 month postoperative/post baseline, 6 months postoperative/post baseline, and 1 year postoperative/post baseline
  Standardized cognitive measure that assesses verbal fluency
Trail Making- Part B | Preoperative/baseline, 1 month postoperative/post baseline, 6 months postoperative/post baseline, and 1 year postoperative/post baseline
  Standardized cognitive measure that assesses executive functioning
Hopkins Verbal Learning Test (HVLT) | Preoperative/baseline, 1 month postoperative/post baseline, 6 months postoperative/post baseline, and 1 year postoperative/post baseline
  Standardized measure to assess new learning and memory
D-KEFS Verbal Fluency Test (FAS) | Preoperative/baseline, 1 month postoperative/post baseline, 6 months postoperative/post baseline, and 1 year postoperative/post baseline
  Standardized measure to assess letter fluency

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Ghogawala, MD, Principal Investigator — Lahey Clinic, Inc.
Locations (3):
- United States (3):
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - University of Buffalo Neurosurgery (UBNS), Buffalo, New York
  - StonyBrook, Stony Brook, New York

REFERENCES:
- [Background] Halliday A, Mansfield A, Marro J, Peto C, Peto R, Potter J, Thomas D; MRC Asymptomatic Carotid Surgery Trial (ACST) Collaborative Group. Prevention of disabling and fatal strokes by successful carotid endarterectomy in patients without recent neurological symptoms: randomised controlled trial. Lancet. 2004 May 8;363(9420):1491-502. doi: 10.1016/S0140-6736(04)16146-1. PMID 15135594
- [Background] Rothwell PM, Goldstein LB. Carotid endarterectomy for asymptomatic carotid stenosis: asymptomatic carotid surgery trial. Stroke. 2004 Oct;35(10):2425-7. doi: 10.1161/01.STR.0000141706.50170.a7. Epub 2004 Aug 26. No abstract available. PMID 15331794